CLINICAL TRIAL: NCT06127355
Title: Gestational Treatment With Ursodeoxycholic Acid Compared to Placebo to Reduce Severity of Gestational Diabetes Mellitus
Brief Title: Gestational Treatment With Ursodeoxycholic Acid Compared to Placebo to Reduce Severity of Gestational Diabetes Mellitus Diagnosed at 24-28 Weeks' Gestation
Acronym: GUARDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMIB-GU-2019-02
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ursodeoxycholic Acid (Experimental): 500 mg of ursodeoxycholic acid (UDCA)
  Interventions: Drug: 500 mg of ursodeoxycholic acid (UDCA)
- Control (Placebo Comparator): 500 mg of Placebo
  Interventions: Other: 500 mg of Placebo

INTERVENTIONS:
Drug: 500 mg of ursodeoxycholic acid (UDCA) — Administration of 500 mg of ursodeoxycholic acid (UDCA) /day
  Arms: Ursodeoxycholic Acid
Other: 500 mg of Placebo — Administration of 500 mg of placebo /day
  Arms: Control

SUMMARY:
The trial will compare the influence of treatment with ursodeoxycholic acid (UDCA) compared to placebo on glycaemic control (primary outcome) in women with GDM after a positive diagnosis at 24-28 weeks of gestation.

The investigators will evaluate maternal and fetal lipid and glucose metabolism. Neonatal health outcomes will also be studied, including the rate of LGA. UDCA is used to treat the commonest liver disease of pregnancy, intrahepatic cholestasis of pregnancy (ICP), and has good safety data to support its use in pregnancy 52-57 ., it means, no studies reported any increase in adverse outcomes associated with UDCA treatment. It is noteworthy that in the largest study 52, 8 serious adverse events were reported, 6 of which were in the placebo group, and none were considered to be related to the trial intervention. There were 72 adverse events: 31 in the ursodeoxycholic acid group and 41 in the placebo group. The same number of patients in each group (n=10) reported adverse events related to gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Women with GDM diagnosed at 24-28 weeks' gestation in accordance with Spanish guidelines in accordance with NDDG criteria, i.e. two or more glucose concentrations (fasting: ≥ 5.8 mmol/L (105 mg/dL), 1 h: ≥10.6 mmol/L, (190 mg/dL) 2 h: ≥9.2 mmol/L (165 mg/dL), 3 h: ≥ 8.1 mmol/L (145 mg/dL)) after a standard 100g OGTT, two fasting blood glucose levels ≥ 126 mg/dl, on different days, or at random ≥ 200 mg/dL or a plasma glucose value greater than 200 mg/dL after OSullivan test
* Planned antenatal care at the same centre (i.e. not planning to move before delivery).
* Singleton pregnancy.
* Informed and written consent.

Exclusion Criteria:

* Age <18 years;
* Multiple pregnancy in current pregnancy;
* Unconscious or very ill;
* Serious mental illness;
* Learning difficulties;
* Not fluent in local language and absence of interpreter.
* Severe congenital anomaly on ultrasound
* Previous diagnosis of diabetes outside of pregnancy
* Significant pre-pregnancy comorbidities that increase risk in pregnancy, for example renal failure, severe liver disease, transplantation, cardiac failure, psychiatric conditions requiring in-patient admission (<1 year)
* Significant co-morbidity in the current pregnancy, nephropathy (estimated GF<60ml/min), other physical or psychological conditions likely to interfere with the conduct of the study and/or interpretation of the trial results
* Participating in another intervention study that will influence the outcome of this trial (to be advised by CI or PI).
* Known allergy/hypersensitivity/intolerance to the active substance or excipients.
* Hypersensitivity to Ursodexosolic acid or to the following excipients: Magnesium stearate, cellulose powder, colloidal silica and sodium carboxymethyl starch, gelatin, titanium dioxide, quinoline yellow, orange yellow S, indigotine.
* Patients with a non-functioning gallbladder, in patients with calcified cholesterol stones, radio-opaque stones, radiolucent gallbladder stones.
* Gastric or duodenal ulcer.
* Liver or intestinal disorders that interfere with the enterohepatic circulation: acute cholecystitis that does not subside, cholangitis, biliary obstruction, pancreatitis due to stones, patients with gastrointestinal-biliary fistula.
* Breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gestational treatment
Enrollment: 113 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Maternal fasting glucose concentration at 36 weeks | Up to 36 weeks
  aiming to maintain all capillary glucose levels between 3.9-7.8mmol/l (70 - 140 mg/dL). The specific pre- and post-meal self-monitored blood glucose (SMBG) targets are ≤5.3mmol/L before breakfast (95 mg/dL), ≤7.8mmol/L 1-hr post meal (140 mg/dL) and ≤6.7mmol/L (120 mg/dL) 2-hr post meal.

SECONDARY OUTCOMES:
Proportion of women requiring insulin treatment | Up to 36 weeks
  Number of women with insuline treatment
Proportion of delivery type | Up to 40 weeks
  Mode of delivery (rates of primary & repeat CS, elective & emergency
Gestational age at delivery, frequency of preterm delivery | Up to 40 weeks
  Age of patient
Infant birth weight | Up to 40 weeks
  Weight in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No